CLINICAL TRIAL: NCT03009968
Title: Reducing Postoperative Catheterization After Urogynecology Surgery: A Randomized Trial
Brief Title: Reducing Postoperative Catheterization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16-2888
Record Dates: First submitted 2017-01-02; First posted 2017-01-04 (Estimated); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Urinary Retention; Urinary Incontinence; Pelvic Organ Prolapse; Urinary Tract Infections
MeSH Terms: conditions — Urinary Retention; Urinary Incontinence; Pelvic Organ Prolapse; Urinary Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional backfill assisted voiding trial (No Intervention): Backfill the bladder with up to 300 ml as tolerated of normal saline or sterile water through an indwelling Foley catheter. The catheter is removed and the patient is given 15 minutes to void and the voided volume is measured. A post void residual (PVR) is measured after voiding (or attempt to void) using either an in and out catheter or a bladder scanner. The participant is considered to have passed the void trial if they have a PVR of less than 100 mL or less than half the voided volume if voided volume is greater than 200 mL.
- Post-void residual free voiding trial (Experimental): The post-void residual free voiding trial (intervention): Backfill the bladder with up to 300 ml as tolerated of normal saline or sterile water through an indwelling Foley catheter. The catheter is removed and the patient is given 15 minutes to void and the voided volume is measured. The participant is considered to have passed the void trial if they void more than 1/2 the instilled volume. A PVR will not be performed.
  Interventions: Other: Post-void residual free voiding trial

INTERVENTIONS:
Other: Post-void residual free voiding trial — Will proceed with voiding trial and assess bladder emptying based on voided amount without checking a post-void residual.
  Arms: Post-void residual free voiding trial

SUMMARY:
After reconstructive pelvic surgery urinary retention occurs in up to 60% of patients requiring an indwelling catheter or self-catheterization (1-5). Up to 35% of women with acute retention experience urinary tract infections in the postoperative period (6, 7). Many women consider being discharged with a Foley catheter to be a surgical complication and describe catheter use as the worst aspect of their surgery(8). At this time there is no consensus within the field of Female Pelvic Medicine and Reconstructive Surgery (FPMRS) on how to best assess voiding function postoperatively. FPMRS providers both within the United States and around the world utilize a variety of void trial methods and varying criteria to determine adequacy of post-operative voiding efficiency (5).

The traditional backfill assisted void trial method involves the assessment of a postvoid residual (PVR) volume obtained either via catheterization or bladder scan (3). Recently, there have been efforts to determine ways to avoid the assessment of a PVR as it is time-consuming and potentially exposes the patient to additional catheterizations (9, 10). Many FPMRS providers utilize the backfill assisted method without assessing a PVR and instead utilize a certain voided volume threshold to determine adequate voiding. However, to date, no one has directly studied this approach or compared the traditional backfill assisted void trial to a PVR-free backfill assisted void trial. By decreasing catheterization and creating a more efficient void trial method, the investigators hope improve patients' postoperative experience and reduce catheterization and risk of urinary tract infection (UTI).

This study aims to compare two void trial methodologies in order to help standardize post-operative care in the urogynecology population. This study also has potential to lead to an overall change in our field and improve the postoperative course for women across the country and abroad.

DETAILED DESCRIPTION:
Data Collection Demographic characteristics (i.e. age, race, body mass index, medical history) will be collected at the time of preoperative visit. On the day of surgery, operative data will be recorded on a standard form to document procedures performed, intra-operative complications (if any), EBL and operative time. Prior to discharge the randomized void trial will be preformed. Data regarding the void trial will be documented on a standard form and will include which void trial was performed, amount backfilled, amount voided, post void residual when assessed, and if the patient was discharged voiding spontaneously, with a Foley catheter or performing CISC. All subjects will be instructed to call our clinical office to report any urinary complaints and treatment for UTI. Information will be collected from electronic medical records regarding any office visits, urine cultures performed or treatment for UTI during this 6-week period. Participants will be called 1 week from the time of surgery to complete the Short-term Catheter Burden Questionnaire.

Pre-operative Visit The preoperative visit may occur up to 3 months prior to surgery. Patients electing to participate in the study will be consented in a private exam to protect confidentiality. Once consented the subjects will be assigned a subject identification number for study identification purposes, which will consist of "A" if the patient's surgery is performed at Rex Hospital or "B" if the patient's surgery is performed at Hillsborough. A number will then follow the letter.

Void Trial Protocols

1. Traditional backfill assisted voiding trial (control): Backfill the bladder with up to 300 ml as tolerated of normal saline or sterile water through an indwelling Foley catheter. The catheter is removed and the patient is given 15 minutes to void and the voided volume is measured. A post void residual (PVR) is measured after voiding (or attempt to void) using either an in and out catheter or a bladder scanner. The participant is considered to have passed the void trial if they have a PVR of less than 100 mL or less than half the voided volume if voided volume is greater than 200 mL.
2. The post-void residual free voiding trial (intervention): Backfill the bladder with up to 300 ml as tolerated of normal saline or sterile water through an indwelling Foley catheter. The catheter is removed and the patient is given 15 minutes to void and the voided volume is measured. The participant is considered to have passed the void trial if they void more than 1/2 the instilled volume. A PVR will not be performed.

If the participant fails the voiding trial through either method they will be discharged to home with an indwelling catheter or with clean intermittent self-catheterization (CISC) per the participants preference. Subjects with an indwelling catheter will return to clinic within 1-3 days for a repeat voiding trial using the same voiding trial guidelines. If the subject is discharged on clean intermittent self-catheterization (CISC) she will document her voided volumes and PVRs at home. Our nurse will then call the participant every 1-2 business days to determine when they can stop CISC (2 consecutive PVRs less than 100 mL). Nurses will document all information into a standardized template in EPIC per routine clinic protocol.

Follow-Up Participants will be scheduled for their post-operative appointment at the time of scheduling their surgery per usual protocol. They will be called 1 week after surgery to complete a questionnaire. The postoperative visit usually takes place approximately 6 weeks after surgery. Any additional visits or calls to Urogynecology clinic prior to their post-operative appointment will be documented in the electronic medical record per routine clinical practice.

All efforts will be made to ensure minimal loss to follow-up of participants. This plan may include efforts such as telephone follow-up or electronic medical record communication with the patient.

Week 1 Phone Call The patient will be called one week after their surgery to answer the questions from the Short-Term Catheter Burden Questionnaire.

Week 6 Visit (-2 weeks/+2 weeks) The primary outcome will be assessed at the time of the post-operative visit with confirmation of need for catheterization. At this visit the subject will also have the patient complete a questionnaire regarding catheter use.

ELIGIBILITY:
Inclusion Criteria:

The study will include women scheduled for pelvic organ prolapse surgery and/or stress urinary incontinence surgery requiring a post-operative voiding trial.

1. 18 years or older
2. English speaking
3. Documented PVR of less than 100mL prior to surgery obtained either during a previous clinic visit or at the time of their preoperative urodynamics evaluation.

Exclusion Criteria:

1. Pregnancy
2. Dependent on catheterization to void preoperatively
3. Patient's undergoing fistula repair, sacral neuromodulation, urethral diverticulum/vaginal mass excision or mesh revision surgery
4. Inability to give informed consent

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-03-17 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Rate of postoperative catheterization | At the time of hospital discharge (0-1 days)
  Rate of postoperative catheterization which is defined as failing the postoperative voiding trial requiring the patients to be discharged to home with a Foley catheter or using clean intermittent self-catheterization (CISC).

SECONDARY OUTCOMES:
Duration of catheterization | From the day of surgery to 6 weeks post op
  The number of days the subjects use either an indwelling Foley catheter or clean intermittent self catheterization starting on day of surgery.
Treatment of clinical-suspected or culture proven urinary tract infection | From the day of surgery to 6 weeks post op
  Antibiotic therapy given for either empiric or culture-proven UTI within the 6 week postoperative period. Any UTI treatment provided within our clinic is routinely documented in the EMR with urine culture results available in laboratory results. Patients will also be instructed to have any records from treatment obtained outside the UNC system to be faxed to our research offices. At the 6 week postoperative visits participants will be asked as well whether they received any antibiotic treatment for UTI during the 6 week postoperative period.
Time spent in the Post Anesthesia Care Unit (PACU). | 0-24 hours
  PACU time will be defined as the time from when the patient leaves the OR and the time the patient is discharged from the PACU. This information is routinely recorded in the EMR by anesthesia and nursing staff. This secondary outcome will only be used in participants who are being discharged to home from the PACU.
Short term catheter burden | 1 week
  Short term catheter burden will be assess using a validated 6-item questionnaire that will be completed 1 week following surgery in patients who failed the post operative voiding trial and are sent home with either indwelling Foley catheter or performing CISC.
Number of post-operative patient calls and subsequent clinic visits. | From the day of surgery to 6 weeks post op
  This will be calculated using electronic medical record documentation and will compare the number of post-operative patient calls and subsequent patient visits between the control and intervention group.

CONTACTS AND LOCATIONS:
Overall Officials: Marcella G Willis-Gray, MD, Principal Investigator — UNC at Chapel Hill, Division of Female Pelvic Medicine and Reconstructive Surgery
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Geller EJ, Hankins KJ, Parnell BA, Robinson BL, Dunivan GC. Diagnostic accuracy of retrograde and spontaneous voiding trials for postoperative voiding dysfunction: a randomized controlled trial. Obstet Gynecol. 2011 Sep;118(3):637-642. doi: 10.1097/AOG.0b013e318229e8dd. PMID 21860294
- [Background] Schiotz HA, Tanbo TG. Postoperative voiding, bacteriuria and urinary tract infection with Foley catheterization after gynecological surgery. Acta Obstet Gynecol Scand. 2006;85(4):476-81. doi: 10.1080/00016340500409877. PMID 16612711
- [Background] Foster RT Sr, Borawski KM, South MM, Weidner AC, Webster GD, Amundsen CL. A randomized, controlled trial evaluating 2 techniques of postoperative bladder testing after transvaginal surgery. Am J Obstet Gynecol. 2007 Dec;197(6):627.e1-4. doi: 10.1016/j.ajog.2007.08.017. PMID 18060956
- [Background] Hakvoort RA, Thijs SD, Bouwmeester FW, Broekman AM, Ruhe IM, Vernooij MM, Burger MP, Emanuel MH, Roovers JP. Comparing clean intermittent catheterisation and transurethral indwelling catheterisation for incomplete voiding after vaginal prolapse surgery: a multicentre randomised trial. BJOG. 2011 Aug;118(9):1055-60. doi: 10.1111/j.1471-0528.2011.02935.x. Epub 2011 Apr 11. PMID 21481147
- [Background] Hakvoort RA, Burger MP, Emanuel MH, Roovers JP. A nationwide survey to measure practice variation of catheterisation management in patients undergoing vaginal prolapse surgery. Int Urogynecol J Pelvic Floor Dysfunct. 2009 Jul;20(7):813-8. doi: 10.1007/s00192-009-0847-4. Epub 2009 Mar 10. PMID 19495543
- [Background] Sutkin G, Alperin M, Meyn L, Wiesenfeld HC, Ellison R, Zyczynski HM. Symptomatic urinary tract infections after surgery for prolapse and/or incontinence. Int Urogynecol J. 2010 Aug;21(8):955-61. doi: 10.1007/s00192-010-1137-x. Epub 2010 Mar 31. PMID 20354678
- [Background] Dieter AA, Amundsen CL, Edenfield AL, Kawasaki A, Levin PJ, Visco AG, Siddiqui NY. Oral antibiotics to prevent postoperative urinary tract infection: a randomized controlled trial. Obstet Gynecol. 2014 Jan;123(1):96-103. doi: 10.1097/AOG.0000000000000024. PMID 24463669
- [Background] Elkadry EA, Kenton KS, FitzGerald MP, Shott S, Brubaker L. Patient-selected goals: a new perspective on surgical outcome. Am J Obstet Gynecol. 2003 Dec;189(6):1551-7; discussion 1557-8. doi: 10.1016/s0002-9378(03)00932-3. PMID 14710061
- [Background] Ingber MS, Vasavada SP, Moore CK, Rackley RR, Firoozi F, Goldman HB. Force of stream after sling therapy: safety and efficacy of rapid discharge care pathway based on subjective patient report. J Urol. 2011 Mar;185(3):993-7. doi: 10.1016/j.juro.2010.10.050. Epub 2011 Jan 19. PMID 21247598
- [Background] Tunitsky-Bitton E, Murphy A, Barber MD, Goldman HB, Vasavada S, Jelovsek JE. Assessment of voiding after sling: a randomized trial of 2 methods of postoperative catheter management after midurethral sling surgery for stress urinary incontinence in women. Am J Obstet Gynecol. 2015 May;212(5):597.e1-9. doi: 10.1016/j.ajog.2014.11.033. Epub 2014 Nov 27. PMID 25434837
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomized trials. Obstet Gynecol. 2010 May;115(5):1063-1070. doi: 10.1097/AOG.0b013e3181d9d421. No abstract available. PMID 20410783
- [Derived] Willis-Gray MG, Wu JM, Field C, Pulliam S, Husk KE, Brueseke TJ, Geller EJ, Connolly A, Dieter AA. Is a Postvoid Residual Necessary? A Randomized Trial of Two Postoperative Voiding Protocols. Female Pelvic Med Reconstr Surg. 2021 Feb 1;27(2):e256-e260. doi: 10.1097/SPV.0000000000000743. PMID 31157716